CLINICAL TRIAL: NCT02872324
Title: Evaluation of the Impact of the Level of Mindfulness on the Management of Patients With Recurrent Depressive Disorders by the Mindfulness Based Cognitive Therapy ( MBCT ): an Exploratory Study
Acronym: MBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-30; 2016-A00691-50 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Patients With Recurrent Depressive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sessions of Mindfulness Based Cognitive Therapy (MBCT) (Experimental)
  Interventions: Other: Procurement questionnaires

INTERVENTIONS:
Other: Procurement questionnaires

SUMMARY:
Mindfulness is both a natural resource of individuals present in all individuals in varying degrees characteristic ability of attention to the experience that unfolds moment by moment without judgment and a practice based on meditation, mindfulness exercises, which aims to enhance two central skills of mindfulness that are the presence and acceptanc. In the context of recurrent depression, the practice of mindfulness meditation in the frame of MBCT is recognized as effective in psychological suffering and relapse. The mechanisms implied in MBCT efficacy are emotional but especially cognitive. Among the cognitive mechanisms, reduction of rumination is a major factor in the action of MBCT, especially for patients with less than three depressive relapses.

This exploratory research focuses on the impact of mindfulness functioning (mindfulness resource level at baseline) on the benefits of MBCT for patients with recurrent depressive disorder.

The objective is to assess whether the level of mindfulness resource of patients with recurrent depression is a factor contributing to the positive effect of a MBCT applied in add-on to conventional care.

This objective will be measured by comparing the clinical improvement of patients secondary to MBCT according to the initial categorization of the mindfulness resource.

Clinical improvement will be more important for patients characterized by a lower initial level of mindfulness resource.

ELIGIBILITY:
Inclusion Criteria:

Major patient Patient with recurrent depression Patient have read, understood and signed the non-opposition form.

Exclusion Criteria:

Inability to understand or read English or French. Individuals unable to personally express their opposition not under whose major legal or private protection of liberty by judicial or administrative decision, or hospital emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Decrease in depression score (Beck Scale) | 24 months
  Decrease in depression score (Beck Scale) after the MBCT program depending on the initial level of full consciousness resource

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Director, Study Director — Assitance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No